CLINICAL TRIAL: NCT06899399
Title: Efficacy and Safety Study of Endovascular Treatment of Asymptomatic Carotid Artery Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Clinical Professor of Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0505400
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Asymptomatic Carotid Artery Stenosis
Keywords: Asymptomatic carotid stenosis; Carotid stenting; Best medical therapy; Randomized controlled trial; Stroke prevention; Endovascular treatment; Carotid artery disease; Ischemic stroke
MeSH Terms: conditions — Carotid Artery Diseases; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal carotid artery stenting and medical treatment (Experimental)
  Interventions: Procedure: Endovascular treatment
- Best Medical Therapy (Active Comparator)
  Interventions: Drug: Best medical treatment

INTERVENTIONS:
Procedure: Endovascular treatment — Participants will receive carotid artery stenting as the primary intervention. The procedure will be performed via femoral artery access (radial access allowed for anatomically challenging cases) with mandatory use of an embolic protection device (EPD). Stent selection and EPD type will be determined by the operator based on lesion characteristics.
  Pre-procedural dual antiplatelet therapy (DAPT: aspirin 100 mg/day + clopidogrel 75 mg/day) will be administered for ≥3-5 days. Post-procedural DAPT will continue for 3 months, transitioning to aspirin monotherapy (100 mg/day) thereafter. Statins and risk factor management (blood pressure、LDL-C, glycemic control) will align with standardized protocols.
  Arms: Internal carotid artery stenting and medical treatment
Drug: Best medical treatment — Participants will receive intensive medical management, including aspirin (75-325 mg/day) or alternative antiplatelet agents (clopidogrel/dipyridamole) for intolerance. Statin therapy and risk factor control targets (blood pressure, lipids, glucose, lifestyle) will mirror the experimental group. Both groups will undergo regular follow-up for adherence monitoring.
  Arms: Best Medical Therapy

SUMMARY:
This study is a multicenter, prospective, open-label, endpoint-blinded, randomized controlled trial designed to evaluate the safety and efficacy of endovascular stenting combined with optimal medical therapy versus optimal medical therapy alone in patients with asymptomatic severe stenosis (70-99%) of the internal carotid artery. The study plans to enroll 982 patients aged 40-80 years who have had no ipsilateral carotid artery-related neurological symptoms in the past six months and who have declined carotid endarterectomy. The primary endpoints include stroke, myocardial infarction, or death within 30 days post-procedure/enrollment, as well as the incidence of ipsilateral stroke from 30 days to one year post-procedure/enrollment. Secondary endpoints include procedural success rate, restenosis rate, changes in cognitive function, and others. The study results will provide high-level evidence-based medical evidence for the treatment selection of patients with asymptomatic carotid artery stenosis.

DETAILED DESCRIPTION:
This multicenter, prospective, open-label, randomized controlled trial with blinded endpoint assessment aims to evaluate the safety and efficacy of endovascular stenting combined with best medical therapy (BMT) versus BMT alone in patients with asymptomatic severe stenosis (70-99%) of the internal carotid artery (ICA). The study will enroll 982 participants aged 40-80 years who have no history of ipsilateral transient ischemic attack (TIA), stroke, or related neurological symptoms within the past 6 months and have declined carotid endarterectomy. The primary objective is to determine whether stenting reduces the composite risk of stroke, myocardial infarction, or death within 30 days post-procedure/enrollment, as well as ipsilateral stroke from 30 days to 1 year. Secondary objectives include assessing procedural success, restenosis rates, cognitive outcomes (measured by Montreal Cognitive Assessment [MoCA] and Mini-Mental State Examination [MMSE]), and long-term clinical outcomes.

The trial will be conducted across multiple centers in China, led by Beijing Tiantan Hospital, Capital Medical University. Participants will be randomly assigned (1:1) via a computer-generated stratified randomization scheme to either the intervention group (endovascular stenting plus BMT) or the control group (BMT alone). BMT includes antiplatelet therapy, lipid-lowering agents, blood pressure control, and management of other cardiocerebrovascular risk factors. Endpoint adjudication will be performed by an independent blinded clinical events committee to minimize bias.

Eligible participants must have severe ICA origin stenosis confirmed by ultrasound, computed tomography angiography (CTA), or digital subtraction angiography (DSA), with contralateral ICA stenosis <70%. Key exclusion criteria include recent symptomatic stenosis, intracranial hemorrhage within 1 year, severe cardiopulmonary comorbidities, contraindications to antiplatelet/anticoagulant therapy, life expectancy <5 years, or anatomical challenges (e.g., Type III aortic arch, severe vascular tortuosity/calcification). Imaging exclusions focus on technical feasibility and safety, such as tandem intracranial stenosis or distal lesions more severe than the target stenosis.

The primary endpoints are the 30-day composite rate of stroke, myocardial infarction, or death, and the incidence of ipsilateral stroke between 30 days and 1 year. Secondary endpoints include technical success (defined as residual stenosis <30% with Thrombolysis in Myocardial Infarction [TIMI] grade 3 flow post-procedure), 30-day and 12-month mortality, restenosis rates, and cognitive changes. Statistical analysis will follow the intention-to-treat principle, with Kaplan-Meier survival analysis and log-rank tests for primary outcomes. Cox proportional hazards models will estimate hazard ratios (HRs) with 95% confidence intervals (CIs). Sensitivity analyses will use per-protocol and as-treated populations.

The study duration is scheduled from August 2024 to July 2028, including a 12-month follow-up period. Ethical approval will be obtained from all participating centers, and the trial will adhere to the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years
2. Severe asymptomatic internal carotid artery stenosis (70-99%) confirmed by ultrasound/CTA/DSA
3. Contralateral ICA stenosis <70%
4. No TIA/stroke related to target lesion in past 6 months
5. Declined carotid endarterectomy
6. Willing to complete 12-month follow-up
7. Signed informed consent by participant/legal representative

Exclusion Criteria:

1. symptomatic internal carotid artery stenosis in the past 6 months
2. Spontaneous intracranial hemorrhage in nearly one year
3. Patients with larger intracranial aneurysms (diameter >5 mm) who cannot undergo prior or concurrent treatment
4. Chronic occlusion without obvious symptoms of cerebral ischemic attack
5. Patients with transient or permanent neurological deficit resulting from Neurological deficits mimicking TIA/stroke from TIA or stroke
6. Common carotid artery ostial lesion
7. Tandem lesions with severe stenosis of the ipsilateral intracranial artery
8. Patients with severe dementia
9. Internal carotid artery dissection
10. Internal carotid artery aneurysm
11. Myocardial infarction within 30 days
12. Ejection fraction <30% or New York Heart Association (NYHA) functional class III or higher; unstable angina, characterized by angina at rest with electrocardiogram changes
13. Cardiogenic embolism, including left ventricular aneurysm, intraluminal filling defects, cardiomyopathy, aortic or mitral valve-prosthetic heart valve, calcified aortic stenosis, infective endocarditis
14. Mitral stenosis, atrial septal defect, atrial septal aneurysm or left chamber myxoma
15. Two or more proximal or main coronary artery stenosis 70%, untreated or recanable
16. Platelets <5 * 104 / uL, INR> 1.5, bleeding time> 1min or heparin-related thrombocytopenia; heparin is a contraindication to antiplatelet drugs; coagulopathy
17. Poor controlled diabetes mellitus, fasting blood glucose> 22 mmol/L and ketone body>+2
18. Malignant tumor or respiratory insufficiency, and a life expectancy of <5 years
19. Severe liver and kidney function impairment, ALT> 3 times the upper limit of normal value or AST> 3 times the upper limit of normal value, blood creatinine increase> 2 times the upper limit of normal value
20. Contrast allergy
21. Other general anesthesia operations are required during the same period
22. Pregnant or lactating women
23. The patient does not attend the clinical trial of other drug or medical device before enrollment
24. The investigator is not considered fit to participate in this clinical study

Imaging exclusion criteria:

1. Type III aortic arch
2. Severe angulation or tortuosity (≥90 degrees) of the common carotid artery or innominate artery that prevents safe and rapid placement of a guiding catheter or long sheath
3. Severe angulation or tortuosity of the internal carotid artery that prevents safe deployment of an embolic protection device or stent. Severe tortuosity is defined as the presence of two or more angles ≥90 degrees within 4 cm of the stenotic lesion
4. Stenosis of the beginning or proximal end of the common carotid artery, innominate artery, distal or intracranial segment of the internal carotid artery, and the stenosis degree is greater than that of the target stenosis
5. The stenotic lesion exhibits severe circumferential calcification, defined as calcification greater than 3 mm in thickness visible in orthogonal views during fluoroscopy. (Note: In elderly subjects aged ≥70 years, anatomical factors such as tortuosity, arch anatomy, and calcification must be assessed more carefully)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint | Within 30 days/ between 30 days and 12 months post-enrollment or post-procedure
  The primary outcome was a composite of any stroke, myocardial infarction (MI), or all-cause mortality within 30 days post-enrollment or post-procedure, plus ipsilateral stroke between 30 days and 12 months post-enrollment/procedure.

SECONDARY OUTCOMES:
Success rate of surgical technique | Surgery completed
  Success rate of surgical technique (defined as final residual stenosis <30%,TIMI grade 3, no dissection or thrombosis after endovascular treatment)
Incidence of myocardial infarction | Within 30 days after surgery or within 30 days of enrollment
  Incidence of myocardial infarction within 30 days after surgery or within 30 days of enrollment
Incidence of ipsilateral stroke | Within 30 days after surgery or within 30 days of enrollment
  Incidence of ipsilateral stroke within 30 days after surgery or within 30 days of enrollment
Incidence of bilateral stroke | Within 30 days after surgery or within 30 days of enrollment
  Incidence of bilateral stroke within 30 days after surgery or within 30 days of enrollment
The incidence of all-cause death | Within 30 days after surgery or within 30 days of enrollment
  The incidence of all-cause death after surgery or within 30 days of enrollment
Cognitive function improvement (MoCA scale) | Within 30 days after surgery or within 30 days of enrollment
  Cognitive function assessment at 30 days after surgery or within 30 days of enrollment (MoCA scale) (optional)
Cognitive improvement (MMSE scale) | 30 days after surgery or within 30 days of enrollment
  Cognitive function assessment (MMSE scale) after surgery or within 30 days of enrollment (optional)
Incidence of ipsilateral stroke | 12 months after surgery or enrollment
  Incidence of ipsilateral stroke at 12 months after surgery or enrollment
The incidence of all-cause death | 12 months after surgery or enrollment
  The incidence of all-cause death at 12 months after surgery or enrollment
Incidence of bilateral stroke | 12 months after surgery or enrollment
  Incidence of bilateral stroke at 12 months after surgery or enrollment
Rate of internal carotid artery restenosis | 12 months after surgery or enrollment
  Rate of internal carotid artery restenosis at 12 months after surgery or enrollment; (Internal carotid artery restenosis definition: Restenosis ≥50% after internal carotid artery stent implantation, peak contraction velocity ratio [PSVR]≥2.0)
Cognitive function improvement (MoCA scale) | 12 months after surgery or within 12 months of enrollment.
  Cognitive function assessment at 12 months after surgery or within 12 months of enrollment (MoCA scale) (optional)
Improvement in cognitive function (MMSE scale) | 12 months after surgery or enrollment
  Improvement in cognitive function (MMSE scale) at 12 months after surgery or enrollment (optional)

CONTACTS AND LOCATIONS:
Overall Officials: Feng Gao, MD, Principal Investigator — Beijing Tiantan Hospital; Zhongrong Miao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No